CLINICAL TRIAL: NCT00741338
Title: A Trial of Antigen-specific Immune Tolerance Induction in Mucopolysaccharidosis I (MPS I) Patients Initiating Enzyme Replacement Therapy With Aldurazyme® (Laronidase)
Brief Title: Immune Tolerance Study With Aldurazyme® (Laronidase)
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Genzyme, a Sanofi Company (Industry)
Collaborators: BioMarin/Genzyme LLC (Industry)
Responsible Party: Sponsor
Organization: Sanofi (Industry)
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ALID02307; 2007-001163-30 (EudraCT Number)
Record Dates: First submitted 2008-08-13; First posted 2008-08-26 (Estimated); Results first posted 2014-07-02 (Estimated); Last update posted 2014-07-02 (Estimated); Status verified 2014-06

CONDITIONS: Mucopolysaccharidosis I
Keywords: MPS I, Mucopolysaccharidosis, Hurler syndrome
MeSH Terms: conditions — Mucopolysaccharidosis I; Mucopolysaccharidoses | interventions — Iduronidase; Cyclosporine; Azathioprine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Cohort 1 (Experimental): Tolerance Induction Period (TIP): Cyclosporine A (CsA) starting at 5 milligram per kilogram (mg/kg) orally three times daily until the target trough concentration of at least 350 nanogram per milliliter (ng/mL) (preferably 400 ng/mL) achieved along with azathioprine (Aza) 2.5 mg/kg/day orally. Once target CsA trough level achieved and maintained for at least 1 week, participants received laronidase 0.058 mg/kg (low-dose) once weekly intravenous (IV) infusion (starting from Day 1) up to Week 12. CsA and Aza were gradually discontinued. Immune Challenge Period (ICP): following TIP, laronidase dose increased to 0.12 mg/kg once weekly IV infusion for 1 week followed by 0.25 mg/kg once weekly IV infusion for 1 week and then 0.58 mg/kg (full-dose) once weekly IV infusion up to Week 39.
  Interventions: Biological: Laronidase; Drug: Cyclosporine A (CsA); Drug: Azathioprine (Aza)
- Cohort 2 (Experimental): TIP: CsA starting at 6.7 mg/kg orally three times daily until the target trough concentration of at least 350 ng/mL (preferably 400 ng/mL) achieved along with Aza 5 mg/kg orally every other day. Once target CsA trough level achieved and maintained for at least 1 week, participants received laronidase 0.058 mg/kg (low-dose) once weekly IV infusion (starting from Day 1) up to Week 18. CsA and Aza were gradually discontinued. ICP: following TIP, laronidase dose increased to 0.12 mg/kg once weekly IV infusion for 1 week followed by 0.25 mg/kg once weekly IV infusion for 1 week and then 0.58 mg/kg (full-dose) once weekly IV infusion up to Week 45.
  Interventions: Biological: Laronidase; Drug: Cyclosporine A (CsA); Drug: Azathioprine (Aza)

INTERVENTIONS:
Biological: Laronidase — 0.058 mg/kg - 0.58 mg/kg IV infusion weekly.
  Other Names: Aldurazyme®
Drug: Cyclosporine A (CsA) — Orally three times daily.
  Other Names: Neoral®
Drug: Azathioprine (Aza) — Orally either every day for Cohort 1 or every other day for Cohort 2.
  Other Names: Imuran®

SUMMARY:
The purpose of this study is to see if treatment with an antigen-specific immunosuppressive can decrease or stop an antibody response to laronidase (Aldurazyme®) during enzyme replacement therapy with laronidase in severe Mucopolysaccharidosis I (MPS I) participants.

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent is required from the parent(s) or legal guardian(s) prior to any protocol-related procedures being performed. (A separate informed consent will be requested from the parent(s) for their genotyping, which is independent of the inclusion)
* Participant's parent(s) or legal guardian(s) allow their child's participation and are willing and able to comply with trial procedures
* The participant must be up to and including 5 years of age at the time of enrollment
* Clinical diagnosis of the severe (Hurler) phenotype of MPS I
* Confirmed presence of 2 nonsense mutations in the alfa-L-iduronidase (IDUA) gene (that is, compound heterozygosity or homozygosity). For the purpose of enrollment, genotyping may be performed by a local laboratory. If no genotyping is performed by a local laboratory, a sample is collected for analysis by a central laboratory before enrollment
* Documented IDUA deficiency with fibroblast, plasma, serum, leukocyte or dried blood spot IDUA enzyme activity assay

Exclusion Criteria:

* The participant has a clinically significant organ disease including: cardiovascular, hepatic, pulmonary, neurologic, or renal disease, other serious intercurrent illness or extenuating circumstances that, in the opinion of the investigator, precludes participation in the trial or potentially decrease survival
* The participant has previously received treatment with laronidase
* The participant has known severe hypersensitivity to any excipients of the delivery solution for laronidase or to any of the other investigational drugs used in the study
* The participant has undergone a haematopoietic stem cell transplant (HSCT), regardless of outcome, or is currently under consideration for such a transplant. If a family later decides to obtain HSCT, the participant will be discontinued from the trial
* The participant has received an investigational product within the 30 days prior to enrollment
* The participant has prior treatment in any experimental protocol (for example, fibroblast injections) that might potentially induce antibodies to laronidase or might affect the interpretation of the participant's antibody response to laronidase
* The participant has received vaccination(s) within 1 month prior to enrollment, or is unwilling to postpone vaccinations during the Tolerance Induction Period in the trial
* The participant is homozygous for thiopurine methyltransferase (TPMT) deficiency, as determined by the genotype (the presence of 2 known null alleles for TPMT) or phenotype (near to complete absence of TPMT enzyme activity)
* The participant has a prior history of tuberculosis or a positive test for latent tuberculosis infection

Max Age: 5 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 7 (Actual)
Dates: Start 2008-09; Primary Completion 2012-09 (Actual); Study Completion 2012-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Genzyme Europe B.V.
Locations (2):
- HCPA, Porto Alegre, Brazil
- Moscow Research Institute for Pediatrics and Children Surgery, Moscow, Russia

REFERENCES:
- [Derived] Giugliani R, Vieira TA, Carvalho CG, Munoz-Rojas MV, Semyachkina AN, Voinova VY, Richards S, Cox GF, Xue Y. Immune tolerance induction for laronidase treatment in mucopolysaccharidosis I. Mol Genet Metab Rep. 2017 Jan 13;10:61-66. doi: 10.1016/j.ymgmr.2017.01.004. eCollection 2017 Mar. PMID 28119821

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study was conducted at 2 centers in Brazil and Russia between September 2008 and September 2013.
Pre-assignment Details: A total of 7 participants were enrolled, 3 in Cohort 1 and 4 in Cohort 2. Of the 4 participants enrolled in Cohort 2, one participant was screen failure.
Period: Overall Study
Arm/Group | Cohort 1 | Cohort 2
Started | 3 | 3
Completed | 3 | 2
Not Completed | 0 | 1
Not completed — Adverse Event | 0 | 1

BASELINE CHARACTERISTICS:
Population: Analysis population included all enrolled participants, including 1 participant who was screen failure.
Groups:
- Total: Total of all reporting groups
Arm/Group | Cohort 1 | Cohort 2 | Total
Number analyzed (Participants) | 3 | 4 | 7
Age, Continuous [Mean (Full Range); unit: years] | 2.60 [1.8 to 3.5] | 3.77 [3.0 to 4.2] | 3.18 [1.8 to 4.2]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 0 | 2
  Male | 1 | 4 | 5

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Who Achieved Immune Tolerance Induction
Description: Immune tolerance induction success was defined as development of an anti-laronidase immunoglobulin G (IgG) antibody titer less than or equal to (<=) 1:3200 after 24 weeks of receiving full-dose (0.58 mg/kg) laronidase therapy.
Time Frame: 24 weeks after start of full-dose laronidase therapy
Population: Safety population included all participants who received any study drug treatment.
Measure: Number; unit: participants
Arm/Group | Cohort 1 | Cohort 2
Number analyzed (Participants) | 3 | 3
participants | 0 | 1

2. Secondary Outcome: Percent Reduction of Urinary Glycosaminoglycan (uGAG) Level From Baseline to the End of Treatment/Early Withdrawal
Description: Urinary Glycosaminoglycan (uGAG) Levels: concentration of glycosaminoglycan (GAG) relative to creatinine in urine. A greater decrease in uGAG level indicates a greater response.
Time Frame: Baseline, end of treatment/early withdrawal (up to 24 weeks after start of full-dose laronidase therapy)
Population: Safety population included all participants who received any study drug treatment.
Measure: Median (Full Range); unit: percent change in uGAG level
Arm/Group | Cohort 1 | Cohort 2
Number analyzed (Participants) | 3 | 3
percent change in uGAG level | -43.80 [-61.70 to -6.70] | -72.50 [-84.20 to -62.50]

ADVERSE EVENTS:
Time Frame: From signature of informed consent up to 30 days after end of treatment/early withdrawal (end of treatment/early withdrawal: up to 24 weeks after start of full-dose laronidase therapy).
Description: Analysis was performed on safety population. In the event a single participant has experienced both a serious and a non-serious form of the same adverse event term, the individual has been included in the numerator ("number of affected participants") of both adverse event tables.
Groups:
- Cohort 2: TIP: CsA starting at 6.7 mg/kg orally three times daily until the target trough concentration of at least 350 ng/mL (preferably 400 ng/mL) achieved along with Aza 5 mg/kg orally every other day. Once target CsA trough level achieved and maintained for at least 1 week, participants received laronidase 0.058 mg/kg (low- dose) once weekly IV infusion (starting from Day 1) up to Week 18. CsA and Aza were gradually discontinued. ICP: following TIP, laronidase dose increased to 0.12 mg/kg once weekly IV infusion for 1 week followed by 0.25 mg/kg once weekly IV infusion for 1 week and then 0.58 mg/kg (full-dose) once weekly IV infusion up to Week 45.
Arm/Group | Cohort 1 | Cohort 2
Serious Adverse Events (participants affected / at risk) | 2/3 | 1/3
Other Adverse Events (participants affected / at risk) | 3/3 | 3/3
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Cohort 1 (N=3) | Cohort 2 (N=3)
Neutropenia (Blood and lymphatic system disorders) | 1 | 0
Bronchopneumonia (Infections and infestations) | 1 | 0
Device related infection (Infections and infestations) | 1 | 0
Respiratory tract infection viral (Infections and infestations) | 0 | 1
Sinusitis (Infections and infestations) | 1 | 0
Bronchospasm (Respiratory, thoracic and mediastinal disorders) | 1 | 0
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Cohort 1 (N=3) | Cohort 2 (N=3)
Anaemia (Blood and lymphatic system disorders) | 0 | 1
Iron deficiency anaemia (Blood and lymphatic system disorders) | 1 | 0
Lymphocytosis (Blood and lymphatic system disorders) | 0 | 1
Neutropenia (Blood and lymphatic system disorders) | 1 | 1
Thrombocytosis (Blood and lymphatic system disorders) | 0 | 1
Abdominal pain (Gastrointestinal disorders) | 2 | 0
Diarrhoea (Gastrointestinal disorders) | 1 | 1
Flatulence (Gastrointestinal disorders) | 0 | 1
Gingival cyst (Gastrointestinal disorders) | 1 | 0
Gingival hyperplasia (Gastrointestinal disorders) | 1 | 0
Nausea (Gastrointestinal disorders) | 1 | 0
Umbilical hernia, obstructive (Gastrointestinal disorders) | 1 | 0
Vomiting (Gastrointestinal disorders) | 1 | 0
Chills (General disorders) | 1 | 0
Hyperthermia (General disorders) | 1 | 1
Influenza like illness (General disorders) | 1 | 0
Medical device complication (General disorders) | 0 | 1
Pyrexia (General disorders) | 2 | 0
Drug hypersensitivity (Immune system disorders) | 1 | 0
Ear infection (Infections and infestations) | 0 | 1
Folliculitis (Infections and infestations) | 1 | 0
Giardiasis (Infections and infestations) | 1 | 0
Gingivitis (Infections and infestations) | 0 | 1
Impetigo (Infections and infestations) | 1 | 0
Laryngitis viral (Infections and infestations) | 1 | 0
Nematodiasis (Infections and infestations) | 1 | 0
Periodontitis (Infections and infestations) | 0 | 2
Rash pustular (Infections and infestations) | 1 | 0
Respiratory tract infection (Infections and infestations) | 0 | 1
Respiratory tract infection viral (Infections and infestations) | 0 | 1
Rhinitis (Infections and infestations) | 0 | 1
Sinusitis (Infections and infestations) | 1 | 0
Upper respiratory tract infection (Infections and infestations) | 3 | 0
Arthropod sting (Injury, poisoning and procedural complications) | 1 | 0
Head injury (Injury, poisoning and procedural complications) | 1 | 0
Blood pressure increased (Investigations) | 0 | 2
Head circumference abnormal (Investigations) | 0 | 1
Red blood cell sedimentation rate increased (Investigations) | 0 | 1
Weight decreased (Investigations) | 0 | 1
Decreased appetite (Metabolism and nutrition disorders) | 1 | 0
Ataxia (Nervous system disorders) | 1 | 0
Anxiety (Psychiatric disorders) | 0 | 1
Bronchospasm (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 2 | 0
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 2 | 0
Stridor (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Alopecia (Skin and subcutaneous tissue disorders) | 1 | 0
Dermatitis allergic (Skin and subcutaneous tissue disorders) | 1 | 0
Dermatitis atopic (Skin and subcutaneous tissue disorders) | 2 | 0
Erythema (Skin and subcutaneous tissue disorders) | 0 | 1
Hand dermatitis (Skin and subcutaneous tissue disorders) | 0 | 1
Heat rash (Skin and subcutaneous tissue disorders) | 1 | 0
Hypertrichosis (Skin and subcutaneous tissue disorders) | 2 | 0
Ingrowing nail (Skin and subcutaneous tissue disorders) | 2 | 0
Papule (Skin and subcutaneous tissue disorders) | 1 | 0
Prurigo (Skin and subcutaneous tissue disorders) | 1 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 0 | 1
Rash (Skin and subcutaneous tissue disorders) | 2 | 0
Rash papular (Skin and subcutaneous tissue disorders) | 1 | 0
Skin maceration (Skin and subcutaneous tissue disorders) | 0 | 1
Urticaria (Skin and subcutaneous tissue disorders) | 1 | 1
Hyperaemia (Vascular disorders) | 1 | 0

LIMITATIONS AND CAVEATS:
Study was discontinued on September 10,2013 due to changing standards of care for this population, practical infeasibility of routinely monitoring plasma CsA in clinical setting, inconclusive results of interim analysis and not due to safety concern.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
If no publication has occurred within 12 months of the completion of the study, the Investigator shall have the right to publish/present independently the results of the study. The Investigator shall provide the Sponsor with a copy of any such presentation/publication for comment at least 30 days before any presentation/submission for publication. If requested by the Sponsor, any presentation/submission shall be delayed up to 90 days, to allow the Sponsor to preserve its proprietary rights.